CLINICAL TRIAL: NCT06446193
Title: A Multi-center, Randomized, Assessor-blind, Superiority, Confirmatory Clinical Trial to Assess Safety and Efficacy of Cognitive Therapy Software 'NDTx-01' for Improving Social Awareness and Interaction in Children and Adolescents With Autism Spectrum Disorder (ASD) or Social Communication Disorder (SCD)
Brief Title: To Evaluate the Efficacy and Safety of 'NDTx-01' in Patients With ASD or SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neudive Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-02; RS-2023-00265178 (Other Grant/Funding Number: Ministry of Health and Welfare, Republic of Korea); B0081112000610 (Other Grant/Funding Number: Daegu-Gyueongbuk Medical Innovation Foundation (KMEDI hub))
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Social Communication Disorder
Keywords: autism spectrum disorder; social communication disorder; digital therapeutics; adolescents; social communication; social skills; social adaptation; autistic; cognitive behavior therapy; social stories; peer relationship; intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Social Communication Disorder; Communication; Social Skills; Social Adjustment; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): NDTx-01 + TAU (Treatment-As-Usual)
  Interventions: Device: NDTx-01; Behavioral: TAU
- The control group (Other): TAU (Treatment-As-Usual)
  Interventions: Behavioral: TAU

INTERVENTIONS:
Device: NDTx-01 — NDTx-01 intervention: Run 'NDTx-01' application on a smartphone 5 times a week, for 6 weeks, 30 sessions in total.
  Arms: The experimental group
Behavioral: TAU — TAU: Autism Spectrum Disorders(ASD) or Social Communication Disorders(SCD)-related treatment/rehabilitation/education

SUMMARY:
The purpose of this study is to demonstrate the superiority of the treatment of cognitive therapy software 'NDTx-01' compared to TAU (Treatment-As-Usual).

DETAILED DESCRIPTION:
This confirmatory clinical trial aims to demonstrate the superiority of 'NDTx-01' by comparing and evaluating the efficacy and safety of the experimental group applying 'NDTx-01' with TAU (Treatment-As-Usual) and the control group applying TAU only.

The study participants will be randomized in a 1:1 as experimental group and control group. The experimental group applies 'NDTx-01' 30 times for 6 weeks (5 times a week) with TAU and the control group gets TAU only. For the primary purpose, the change in the adaptive behavior combination (ABC) score of the Korean version of the Vineland Adaptive Behavior Scale-II (K-VABS-II) at 42 days compared to the baseline will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between the ages of 10 and 18
* Diagnosed with autism spectrum disorder (ASD) or social communication disorder (SCD) based on the clinical judgment of a psychiatrist according to DSM-5 diagnostic criteria
* Participants who are able to install 'NDTx-01' on an Android smartphone and use it alone or with the help of their guardian
* Participants who are able to comply with the recommended application time for the investigational medical device (6 weeks, 30 times, 5 times a week)
* Participants who have agreed not to use any other medical devices besides the investigational medical device during the clinical trial
* Participants who agree that there should be no change in the use of drugs which can significantly affect one's sociality during the clinical trial (If there is a drug being taken during screening, it can be taken continuously, but the total daily dose, ingredients, etc., should remain unchanged until the end of the study visit.)
* Participants who agree not to participate in other Applied Behavior Analysis (ABA) treatment/rehabilitation/education, social treatment/rehabilitation/education program (If there is treatment/rehabilitation/education being received during screening, it can be received continuously, but the number of applications and treatment methods should remain unchanged until the end of the study visit.)
* Participants who and whose parents (legal guardians) have volunteered to participate in this clinical trial and have given written consent to the subject description and consent form
* Participants willing to comply with the clinical trial procedures

Exclusion Criteria:

* A risk of clinically significant behavioral problems, emotion regulation problems, psychotic symptoms, self-harm, or other harm at a level that affects the treatment process
* Severe acute/chronic medical or mental illness
* Serious trauma or surgery performed within 4 weeks before the screening date
* Participants with other disabilities such as severe neurological diseases (e.g. brain lesions, mental disorders, etc.)
* Participants who are currently participating in another clinical trial or have participated in another clinical trial within 30 days before the screening date
* Participants with a previous history of using NDTx-01, the investigational device
* Participants who have a change in the usage or dosage of drugs which can significantly affect one's sociality, or a change in participation in treatment/rehabilitation/education programs that can significantly affect one's sociality within 8 weeks before the baseline date of the clinical trial
* In other cases where the investigator determines that participation in the clinical trial is inappropriate due to ethical reasons or the possibility of influencing the results of the clinical trial

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Adaptive Behavior Composite score of K-VABS-II (Korean Vineland Adaptive Behavior Scales-Ⅱ) at Day 42 | Baseline, Day 42
  The K-VABS-II is a tool used to assess adaptive behavior and functioning in individuals from birth to 99 years old. It evaluates personal and social skills necessary for everyday living. The scores (standard scores) range from 55 to 145, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Change from Baseline in Adaptive Behavior Composite score of K-VABS-II (Korean Vineland Adaptive Behavior Scales-Ⅱ) at Day 28 | Baseline, Day 28
  The K-VABS-II is a tool used to assess adaptive behavior and functioning in individuals from birth to 99 years old. It evaluates personal and social skills necessary for everyday living. The scores (standard scores) range from 55 to 145, with higher scores indicating better outcomes.
Change from Baseline in K-VABS-II (Korean Vineland Adaptive Behavior Scales-Ⅱ) at Day 28 and Day 42 | Baseline, Day 28, Day 42
  The K-VABS-II is a tool used to assess adaptive behavior and functioning in individuals from birth to 99 years old. It evaluates personal and social skills necessary for everyday living. The scores (standard scores) range from 55 to 145, with higher scores indicating better outcomes.
Change from Baseline in SRS-2 (Korean Social Responsiveness Scale-2) at Day 28 and Day 42 | Baseline, Day 28, Day 42
  The SRS-2 consists of a series of questions answered by parents or caregivers who observe the individual's behavior. It is a tool used to assess social skills, social cognition, and behaviors associated with autism spectrum disorders (ASD) in children and adolescents. It's designed to help clinicians, educators, and researchers identify and understand social impairments commonly seen in individuals with ASD or other developmental disorders. The T scores range from 34 to 128, with higher scores indicating worse outcomes.
Change from Baseline in K-PRQ-CA (Korean Parenting Relationship Questionnaire - Child & Adolescent) at Day 28 and Day 42 | Baseline, Day 28, Day 42
  The K-PRQ-CA is a tool designed to assess the quality of the relationship between parents and their children or adolescents. It's used to evaluate various aspects of the parent-child relationship, including communication, support, discipline, and overall satisfaction. The T scores of K-PRQ-CA are estimated to be 20 to 80 (T score mean 50, standard deviation 10), with higher scores indicating better outcomes.
Change from Baseline in KIPR (Korean Inventory of Peer Relationships) at Day 28 and Day 42 | Baseline, Day 28, Day 42
  The KIPR is a tool used to assess peer relationships among Korean children and adolescents. It's designed to measure various aspects of peer interactions, including social skills, peer acceptance, peer rejection, and the quality of friendships. The T scores of KIPR are estimated to be 20 to 80 (T score mean 50, standard deviation 10), with higher scores indicating worse outcomes.
Change from Baseline in EQ-5D-5L (EuroQol Five Dimension Five Level Scale) at Day 42 | Baseline, Day 42
  The EQ-5D-5L is a standardized measure of health-related quality of life developed by the EuroQol Group. It's used to assess a person's health status and well-being across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The "5L" in EQ-5D-5L stands for "five levels," indicating that each dimension has five response levels ranging from no problems to extreme problems. The score for each dimension is from 1 to 5, with higher scores indicating worse outcomes. And the score ranging from 0 to 100 means that the higher the score, the better the outcome.
Change from Baseline in CGI-S (Clinical Global Impression-Severity) at Day 28 and Day 42 | Baseline, Day 28, Day 42
  The CGI-S is a widely used clinician-rated scale designed to assess the overall severity of a patient's condition in clinical trials. Clinicians typically rate the CGI-S on a seven-point scale, where each point represents a different level of severity. The score ranges from 1 to 7, with higher scores indicating worse outcomes.
CGI-I (Clinical Global Impression-Improvement) at Day 28 and Day 42 | Day 28, Day 42
  The CGI-I is a clinician-rated scale used to assess changes in a patient's overall clinical condition or improvement over time, particularly in clinical trials. Clinicians typically rate the CGI-I on a seven-point scale, where each point represents a different level of improvement compared to baseline. The score ranges from 1 to 7, with higher scores indicating worse outcomes.
NDTx-01 Satisfaction Questionnaire at Day 42 | Day 42
  The 'NDTx-01 Satisfaction Questionnaire' includes 4 questions related to satisfaction with the experience of using the investigational device. The score for each question is from 0 to 10, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Sook Joung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Daegu Catholic University Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No